CLINICAL TRIAL: NCT02315092
Title: Evaluation of Fluorescence-image Guided Wound Assessment vs. Standard Practice
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Judy Dan Research and Treatment Centre (Unknown)
Responsible Party: Principal Investigator, Ralph DaCosta, Scientist, University Health Network, Toronto
Other Study IDs: 14-8303
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Foot Ulcer, Diabetic; Bacteria
Keywords: Diabetic Foot Ulcers; Bacteria; Fluorescence
MeSH Terms: conditions — Diabetic Foot | interventions — Optical Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiological samples (skin and wound swabs)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic foot ulcers: Patients who present with diabetic foot ulcers will undergo fluorescence imaging.
  Interventions: Device: Fluorescence Imaging

INTERVENTIONS:
Device: Fluorescence Imaging — Wounds will be imaged using violet light (405 nm) illumination to locate areas with bacterial presence to guide swabbing.

SUMMARY:
The current trial aims to compare the assessment of diabetic foot ulcers by fluorescence image guidance to standard practice. The device will be used to acquire fluorescence images of diabetic foot ulcers: when wounds are illuminated by violet/blue light, most pathogenic bacterial species emit a unique red fluorescence signal. The device is intended to be used as part of the clinical assessment process, which may include visual assessment, signs of heat or high temperature, the presence of exudate, and redness in the area. Images will guide the clinician to inspect, sample or further evaluate areas where fluorescing bacteria is present. This study will allow us to determine the benefit of fluorescence image-guided procedure as compared to standard clinical practice to assess bacterial burden in diabetic foot ulcers. Microbiological swabbing under standard practice and fluoresce-guided imaging will be performed in order to compare the two techniques.

DETAILED DESCRIPTION:
Chronic wounds and their associated care are a burden to patients and health care systems worldwide. Microbiological testing of wound samples is often used to identify and quantify bacterial species, the latter of which may be both an objective quantitative indicator of infection and a predictive correlate of healing. Microbiology reports contain useful information about microbial identities, antibiotic susceptibility, and semi-quantitative bacterial growth rates, but these data typically represent the bacterial load in the wound centre only, and often arrive 3-5 days later. There is an unmet clinical need to improve the microbiological sampling and treatment of wound infections. To address this need, we developed a handheld portable imaging device that obtains white light (WL) and fluorescence (FL) images (or video) of normal skin and wounds in high-resolution and in real-time, which can be used at the point-of-care. It was demonstrated in previous studies that the device1) provides image-guidance for tissue sampling, detecting clinically-significant levels of pathogenic bacteria and wound infection otherwise overlooked by conventional sampling and 2) provides image-guidance for wound treatment, accelerating wound closure compared with conventional therapies and quantitatively tracking long-term changes in bacterial bioburden and distribution in wounds.

The current trial aims to compare the assessment of diabetic foot ulcers by fluorescence image guidance to standard practice. The device will be used to acquire fluorescence images of diabetic foot ulcers: when wounds are illuminated by violet/blue light, most pathogenic bacterial species emit a unique red fluorescence signal. The device is intended to be used as part of the clinical assessment process, which may include visual assessment, signs of heat or high temperature, the presence of exudate, and redness in the area. Images will guide the clinician to inspect, sample or further evaluate areas where fluorescing bacteria is present. This study will allow us to determine the benefit of fluorescence image-guided procedure as compared to standard clinical practice to assess bacterial burden in diabetic foot ulcers. Microbiological swabbing under standard practice and fluoresce-guided imaging will be performed in order to compare the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who present with a diabetic foot ulcer and are receiving standard wound care treatment.
* 18 years and older

Exclusion Criteria:

* Treatment with an investigational drug within 1 month before study enrolment
* Inability to consent
* Any contra-indication to routine wound care and/or monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with a diabetic foot ulcer and are receiving standard wound care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlation of localized fluorescence signals in acquired images with microbiological samples | At study visit (only one study visit)
  Microbiological swabs will be taking from fluorescence positive regions to correlate with bacterial presence
Comparison of number/variety of bacteria obtained by fluorescence-guided sampling vs. standard practice | At study visit (only one study visit)
  Microbiological swabs will be taking from the wound using standard practice and following fluorescence-image guidance

SECONDARY OUTCOMES:
Assessment of the clinical functionality of the K2 Imaging Device | At study visit (only one study visit)
  Users feedback

CONTACTS AND LOCATIONS:
Overall Officials: Ralph S DaCosta, PhD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Judy Dan Research and Treatment Centre, Toronto, Ontario, Canada